CLINICAL TRIAL: NCT03434613
Title: A Randomized, Prospective, Open Label, Active Control, Phase IV Study to Evaluate the Effects of Statin Monotherapy or Statin / Ezetimibe Combination Therapy on Hepatic Steatosis in Patients With Hyperlipidemia and Nonalcoholic Fatty Liver Disease
Brief Title: Phase IV Study to Evaluate the Effects of Statin Monotherapy or Statin / Ezetimibe Combination Therapy on Hepatic Steatosis in Patients With Hyperlipidemia and Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-1168
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Nonalcoholic Fatty Liver Disease; Dyslipidemias
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This study will conduct to evaluate the efficacy of liver fat lowering and safety of rosuvastatin 5mg alone or in combination with rosuvastatin 5mg / ezetimibe 10mg for 6 months.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin monotherapy (Active Comparator): Rosuvastatin 5mg 1T daily for 6 months
  Interventions: Drug: Rosuvastatin
- Rosuvastatin + ezetimibe combination therapy (Experimental): Rosuvastatin 5mg / Ezetimibe 10mg combination 1T daily for 6 months
  Interventions: Drug: Rosuvastatin/ezetimibe combination

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 5mg 1T daily for 6 months
  Arms: Rosuvastatin monotherapy
Drug: Rosuvastatin/ezetimibe combination — Rosuvastatin 5mg / Ezetimibe 10mg combination 1T daily for 6 months
  Arms: Rosuvastatin + ezetimibe combination therapy

SUMMARY:
To investigate the therapeutic effect of ezetimibe on nonalcoholic fatty liver disease, the effect of rosuvastatin 5mg monotherapy and rosuvastatin 5mg / ezetimibe 10mg combination therapy n patients with hyperlipidemia and fatty liver will be compared and analyzed.

This study included a total of 70 patients (35 per subgroup) for randomized controlled trials with prospective, open label, randomized, single-institution clinical trials.

The drug will be maintained for a total of six months. The primary endpoint is the difference of liver fat change measured by MRI-PDFF in colocalized regions of interest within nine liver segments between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 19 and over, under 80 years of age
* Patients diagnosed with fatty liver by abdominal ultrasonography or liver fibroscan. (In case of patients who were diagnosed fatty liver by liver scan, we will conduct abdominal ultrasonography for screening purposes)
* In the Domestic Dyslipidemia Treatment Guideline, patients with hyperlipidemia A. LDL-C is more than 130mg / dL when there is less than 1 major risk factor B. LDL-C 100 mg / dL or more if there are two or more major risk factors C. High-risk patients with carotid stenosis> 50%, abdominal aortic aneurysm, and diabetes mellitus had LDL-C> 70 mg / dL

D. The main risk factors are as follows:

i. smoking ii. Hypertension - systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg or antihypertensive iii. Low HDL cholesterol (<40 mg / dL) iv. Age - Male 45+, Female 55+ v. Family history of early onset coronary artery disease - Parents, siblings with a history of coronary artery disease in men under 55 and women under 65 vi. High HDL cholesterol (60 mg / dL) or more is regarded as a protective factor and one of the total risk factors is reduced

* Even if it does not meet the criteria for hyperlipidemia, it is possible to select the subject when there is evidence of atherosclerosis on the test (carotid ultrasonography etc)
* Those who already use statin as a treatment for hyperlipemia should participate after a washout period of 1-2 weeks.
* Controlled diabetic patients (HbA1c ≤9.0%), no change in type of oral or injectable hypoglycemic agents for the last 12 weeks
* Those who voluntarily agreed to participate in clinical trials after hearing the explanation of the clinical trial
* Those who understand the content of the clinical trial and are able to participate in the trial by the end of the clinical trial

Exclusion Criteria:

* Diabetic patients other than type 2 diabetes, including type 1 diabetes and gestational diabetes
* Those who have a previous history of medication with ezetimibe or discontinuation due to side effects after medication
* Patients who have had a history of discontinuation of statin therapy due to side effects after medication,
* Unregulated diabetic patients (those who have changed the type of oral or injectable hypoglycemic agent within 12 weeks prior to Visit 1 or who have HbA1c> 9.0% at screening time (Visit 1)
* patients with acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma, and patients with a history of ketonic acidosis (within 6 months)
* Those who use thiazolidinedione and SGLT2i drugs which can affect fatty liver as a diabetes treatment drug
* Patients who meet the criteria for alcoholism in fatty liver disease (210 g / week for men in the last two years, 140 g / week for women)
* Chronic liver disease (including hemochromatosis, liver cancer, autoimmune liver disease, Child-Pugh score> 7points, platelet <75,000mm2, prothrombin time> 16s), viral hepatitis -A, B,
* People who take drugs that can cause fatty liver (amiodarone, methotrexate, tamoxifen, valproate, corticosteroids, etc.)
* Patients who are allergic or hypersensitive to the drug or its constituents
* Patients who were treated with oral or parenteral corticosteroids chronic (within consecutive 14 days) within 8 weeks before screening
* Patients with genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder
* Patients with malnutrition, starvation, weakness (including severe infections, pre- and post-operative trauma patients), pituitary dysfunction or adrenal insufficiency
* Serum levels of alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase are increased over 5-fold elevation of the normal range upper limit [ULN] or 5-fold elevation of the serum total bilirubin level. )
* Currently taking medication for weight loss
* Patients with a history of malignant tumors within the past 2 years or malignant tumors that are currently undergoing treatment or progression
* Patients with a history of substance abuse or alcohol intoxication within 12 weeks
* Human immunodeficiency virus (HIV)
* Patients with severe infection, pre- and post-operative, and severe trauma
* Patients with acute cardiovascular disease within 12 weeks (patients with unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass grafting, or coronary intervention)
* Patients with renal failure, chronic renal disease (estimated glomerular filtration rate <60 mL / min / 1.73 m2)
* Anemic patients with a Hb level of less than 10.5 g / dl
* Surgical or medical conditions that may affect the absorption, distribution, metabolism and excretion of a drug, including, but not limited to, gastrectomy, gastroenterostomy, History of major gastrointestinal surgery such as small bowel resection, gastrointestinal bypass, gastrointestinal stapling, current active gastritis, gastrointestinal / rectal bleeding, active inflammatory bowel syndrome within the last 12 months, etc.
* Pregnant or lactating women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
liver fat change measured by MRI-PDFF in colocalized regions of interest within each of nine liver segments | 6 months
  MRI is used to measure the fat fraction in 9 liver segments, and this test has been reported to be more sensitive than the biopsy-based steatosis grade assessment in confirming liver fat changes in previous studies

SECONDARY OUTCOMES:
Liver fibrosis measured by MRE(magnetic resonance elastography) | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: Liver fibrosis measured by magnetic resonance elastography
Change in hepatic steatosis index - controlled attenuation parameter (CAP) | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: controlled attenuation parameter (CAP)
Change in hepatic fibrosis index - liver stiffness measurement (LSM) measured by transient liver elastography (Fibroscan®; Echosens, Paris, France) | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: liver stiffness measurement (LSM) measured by fibroscan
Changes in body weight (kg) before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: body weight
Changes in waist circumference (cm) before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: WC
Changes in systolic & diastolic blood pressure (mmHg) before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: SBP, DBP
Changes in serum concentrations of insulin (µU/mL), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: fasting insulin
Changes in serum concentrations of fasting glucose (mg/dL), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: fasting glucose
Changes in serum concentrations of HbA1c (percent), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: HbA1c
Change in insulin sensitivity determined by homeostatic model assessment insulin resistance (HOMA-IR) and beta cell function determined by HOMA-beta | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: HOMAIR, HOMA-beta
Changes in serum concentrations of free fatty acid (μEq/L), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: free fatty acid
Changes in serum concentrations of platelet (×103/ μL), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: platelet
Changes in serum concentrations of alkaline phosphate (U/L) and gamma-GT(U/L), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: Alk,phos, GGT
Changes in serum concentrations of total bilirubin (mg/dL), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: total bilirubin
Changes in serum concentrations of liver enzymes (aspartate aminotransferase and alanine aminotransferase (IU/L)), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: ALT, AST
Changes in serum lipids (total cholesterol, triglyceride, HDL cholesterol, and LDL cholesterol (mg/dL)), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: LDL-C, TG, HDL, TC
Changes in serum concentrations of CRP (mg/dL), before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: High-sensitivity CRP
Changes in the level of liver injury markers including IL-1beta, IL-8, IL-18 (pg/mL) before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: biomarker ( IL-1b, IL-8, IL18)
Changes in plasminogen activator inhibitor-1 (ng/mL) in peripheral blood mononuclear cells, before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: tPAI-1
Changes in BMI (kg/m^2) before and after the administration of rosuvastatin with/without ezetimibe | 6 months
  The secondary endpoint is to analyze the changes before and after drug administration for the following items: BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of Internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loomba R, Sirlin CB, Ang B, Bettencourt R, Jain R, Salotti J, Soaft L, Hooker J, Kono Y, Bhatt A, Hernandez L, Nguyen P, Noureddin M, Haufe W, Hooker C, Yin M, Ehman R, Lin GY, Valasek MA, Brenner DA, Richards L; San Diego Integrated NAFLD Research Consortium (SINC). Ezetimibe for the treatment of nonalcoholic steatohepatitis: assessment by novel magnetic resonance imaging and magnetic resonance elastography in a randomized trial (MOZART trial). Hepatology. 2015 Apr;61(4):1239-50. doi: 10.1002/hep.27647. Epub 2015 Feb 27. PMID 25482832
- [Derived] Cho Y, Rhee H, Kim YE, Lee M, Lee BW, Kang ES, Cha BS, Choi JY, Lee YH. Ezetimibe combination therapy with statin for non-alcoholic fatty liver disease: an open-label randomized controlled trial (ESSENTIAL study). BMC Med. 2022 Mar 21;20(1):93. doi: 10.1186/s12916-022-02288-2. PMID 35307033